CLINICAL TRIAL: NCT00907686
Title: Prevention of Transfusion-transmitted CMV (TT-CMV) in Lowbirth Weight Infants (LBWI; ≤1500 Grams) Using CMV Seronegative and Leukoreduced Transfusions.
Brief Title: TT-CMV Observational Birth Cohort Study
Acronym: TT-CMV
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Cassandra D Josephson, Associate Professor, Emory University
Other Study IDs: IRB00014684; P01HL086773-01A1 (NIH); NCT00907686 (Other: Clinical Trials.gov)
Record Dates: First submitted 2009-05-21; First posted 2009-05-22 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Cytomegalovirus Disease
Keywords: Transfusion Transmitted Cytomegalovirus (TT-CMV); Low birthweight infants (LBWIs); Leukoreduction and filter failure; CMV Seronegative blood products
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole Blood, Urine, Breast Milk
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- LBWIs of CMV-positive mother: LBWIs born to CMV-positive mothers
- CMV Sero-negative & Sero-postive LBWIs: LBWIs of CMV sero-negative & sero-positive mothers

SUMMARY:
The spread of viruses through transfusions is the cause of serious illness and death in recipients whose immune systems are unable to fight infection. Another group of patients whose immune systems are underdeveloped and can be affected by a particular virus known as cytomegalovirus (CMV) is low birthweight infants (LBWIs). CMV can be spread through the placenta, during the birth process, through breast milk, while in the hospital or while caring for someone carrying the virus as well as through a transfusion, known as transfusion-transmitted (TT-CMV).

The spread of TT-CMV in LBWIs can be curtailed by transfusing blood products that are CMV negative as well as to filter the white cells in blood that carry the virus (leukoreduction). The purpose of this study is to see if the use of these two strategies can lower the spread of CMV through a transfusion. How "safe" the blood actually is through leukoreduction is not known and CMV still occurs in LBWIs. It is not clear whether this approach is optimal or whether additional safety steps are needed to completely prevent TT-CMV. Specific actions that could tell us when virus has reached the blood product or breast milk is to test each of these to determine if virus slipped "unnoticed" and/or when the product was not thoroughly filtered.

In this study, the investigators believe that the use of both prevention strategies will result in a lower rate of TT-CMV, and that the "cause" of TT-CMV may be found in the presence of CMV at the DNA level or by unfiltered white cells that remain in the blood product. Thus, the most significant clinical question that remains to be addressed is whether this double strategy for transfusion safety actually provides a "zero CMV-risk" blood supply or whether further safety measures (DNA testing + 100% leukoreduction) must be used to protect this extremely vulnerable patient group from CMV infection. This birth cohort study will be done with 6 participating NICUs, and will study both CMV positive and negative mothers in order to estimate the rate and pathway of CMV transmission to the LBWI who receives a transfusion. Another study goal is to compare or link any CMV infection by either transfused units where the virus was undetected, or filter failure. If CMV disease occurs, the investigators will be able to describe the course and outcome in LBWIs who develop TT-CMV.

DETAILED DESCRIPTION:
The primary aim of this birth cohort study is to estimate the incidence of TT-CMV in LBWIs who receive a combination of CMV-seronegative + leukoreduced blood products. That is to say, the effectiveness of the two strategies coupled together will be assessed in the prevention of TT-CMV in at-risk LBWI born to CMV-negative and CMV-positive mothers.

The following hypothesis relates to this primary aim, that the incidence of TT-CMV is elevated in the population of LBWIs born the CMV-positive mothers. According to reports in the literature, breakthrough TT-CMV infection will occur at low rates (< 2.5% incidence) in LBWIs of CMV-negative mothers transfused with seronegative plus leukoreduced blood components.

The secondary aim of this study is to detect CMV DNA and/or elevated residual WBC counts in blood components transfused to LBWIs and to determine whether these results are related to episodes of breakthrough TT-CMV in this study population.

Original sample size considerations were based on estimating and comparing the rates of TT-CMV infection in VLBW infants born to CMV-seropositive mothers or CMV-seronegative mothers. Assuming a 2.55% TT-CMV rate for infants born to CMV-seropositive mothers and a 0.5% TT-CMV rate for infants born to CMV-seronegative mothers, a sample size of 650 infants per group would need to be recruited to detect a difference of approximately 2% in the TT-CMV rate with 80% power (2-sided Fisher's exact test at the 5% significance level).

After three years of accrual and follow-up the incidence of TT-CMV was 0%. Sample size calculations were revised using a 95% confidence interval for a single group of VLBW infants regardless of maternal CMV serostatus. The necessary sample size was 300 transfused VLBW infants based on a one-sided exact 95% confidence interval for a single proportion of 0.0 with an upper bound of 0.01.

ELIGIBILITY:
Inclusion Criteria:

* All LBWIs whose weight is ≤ 1500 grams at birth
* LBWI is within first five days of life

Exclusion Criteria:

* LBWI not expected to live past first seven days of life
* LBWI has a severe congenital abnormality
* LBWI has received a RBC or platelet transfusion at another institution prior to transfer
* LBWI has received an in-utero transfusion
* LBWI is clinically suspected of having toxoplasmosis, rubella, herpes infection(s) at birth
* Refusal by the mother to grant consent for herself and/or refusal to grant consent for her LBWI
* If the mother of the child has previously participated in this study

Ages: 1 Hour to 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Low birthweight infants in NICU.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2010-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Estimate the incidence of TT-CMV in LBWIs who receive CMV-seronegative plus leukoreduced blood products. | 90 days study observation
  The effectiveness of these two strategies coupled together will be assessed in the prevention of TT-CMV in at-risk LBWI born to CMV-negative and CMV-positive mothers.

CONTACTS AND LOCATIONS:
Overall Officials: Cassandra Josephson, MD, Study Director — Emory University
Locations (3):
- United States (3):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia

REFERENCES:
- [Derived] Josephson CD, Caliendo AM, Easley KA, Knezevic A, Shenvi N, Hinkes MT, Patel RM, Hillyer CD, Roback JD. Blood transfusion and breast milk transmission of cytomegalovirus in very low-birth-weight infants: a prospective cohort study. JAMA Pediatr. 2014 Nov;168(11):1054-62. doi: 10.1001/jamapediatrics.2014.1360. PMID 25243446
- [Derived] Josephson CD, Castillejo MI, Caliendo AM, Waller EK, Zimring J, Easley KA, Kutner M, Hillyer CD, Roback JD. Prevention of transfusion-transmitted cytomegalovirus in low-birth weight infants (</=1500 g) using cytomegalovirus-seronegative and leukoreduced transfusions. Transfus Med Rev. 2011 Apr;25(2):125-32. doi: 10.1016/j.tmrv.2010.11.004. Epub 2011 Feb 23. PMID 21345642